CLINICAL TRIAL: NCT03725813
Title: Person-centred Inpatient Care - a Quasi-experimental Study Within an Internal Medicine Context
Brief Title: Study Evaluating the Effect of Person-centred Care for Patients Admitted for Inpatient Care at an Internal Medicine Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Person-centred care
Record Dates: First submitted 2018-10-16; First posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Endocrine System Diseases; Gastrointestinal Diseases
Keywords: Person-centred care; Intervention; Inpatient care; Satisfaction of care; quasi-experimental; internal medicine
MeSH Terms: conditions — Endocrine System Diseases; Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: A quasi- experimental study with non-equivalent control group design, pretest-posttest study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Person-centred inpatient care (Experimental): Person-centred inpatient care
  Interventions: Other: Person-centred inpatient care

INTERVENTIONS:
Other: Person-centred inpatient care — The intervention comprises three sequential steps in the care process. The first two steps follow one after the other in conjunction with admission to the ward: 1) person-centred assessment, and 2) creation of a person-centred health plan. Persistent person-centred inpatient care, the third step, is practiced throughout the hospital stay, and is a component of the quality and patient safety program.
  The model is systematically applied to all patients admitted to the unit. All staff are trained in PCC before implementation of the intervention.

SUMMARY:
Patients admitted to internal medicine care environments have complex care needs and must be treated as persons with resources and responsibilities. Person-centred care is defined as care in which the caregiver aims to get to know the patient as a person, and the care comprises a holistic approach to assess patients' needs and resources. There is strong motivation for future health care to transform into an approach that acknowledges and endorses every patient's resources, interests and needs. There is limited existing research on the benefit of implementing person-centred care in internal medicine care environments for all patients regardless of diagnosis or care pathway. Little is known about the effects of person-centred inpatient care on patients' satisfaction with care. This study includes adult patients admitted to an internal medicine inpatient unit regardless of reason for admission. The aim of the study is to evaluate effects of person-centred inpatient care on care processes, in terms of satisfaction with care and person-centred content in medical records and to evaluate effects on self-reported health and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* acute or elective admission with a minimum projected in-hospital stay of 24 hours
* age ≥ 18 years
* conscious and alert, with no delay in response.

Exclusion Criteria:

* cognitive impairment or a judgment by the caregivers that inclusion was not in the best interests of the patient (e.g. end of life care, impaired psychological wellbeing).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Satisfaction with care comprise patients' evaluations of caregivers' identity-oriented approach and the sociocultural atmosphere at the ward. | From date of admission until the date of discharge, up to 60 days of hospitalization.
  The outcome is assessed with the questionnaire Quality from the Patient Perspective. The questionnaire comprises four dimension of with two dimensions is used: Identity-oriented approach (13 items) and the sociocultural atmosphere (5 items). One item from the medical competence subscale (effective pain relief) and one additional item on provision of information about medications is also used. Two kinds of assessments are being made at each item: whether things were being done (perceived reality) and whether the right things were being done (subjective significance). For the primary outcome only the assessments of perceived reality are being used. Items are rated on a four-point response scale ranging from 1 (do not agree at all) to 4 (completely agree). Each item also has a response option of "not applicable". Subscales can be reported item by item or combined in a subscale score (average of all responses within the subscale).
Person-centred content in medical records | From date of admission until the date of discharge, up to 60 days of hospitalization.
  Degree of person-centredness in medical records

SECONDARY OUTCOMES:
Self-reported health assessed with EQ-5D-5L | at the date of discharge, an average of 5 days after inclusion
  Self-reported health is measured with the EuroQual-5Dimensions-5Levels questionnaire (EQ- 5D- 5L). The questionnaire comprises 1 item per dimension. The dimensions of importance for health which are included are; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Patients rate each item on a scale ranging from 1 (no problems) to 5 (extreme problems/unable to). A unique health state is defined by combining 1 level from each of the 5 dimensions. The questionnaire also includes EQ-VAS, in which the patients grade their current health status on an analogue scale from 0 (worst health) to 100 (best health).
Physical and psychological wellbeing assessed with the Quality from the Patient Perspective questionnaire | at the date of discharge, an average of 5 days after inclusion
  Patients rated their physical and psychological wellbeing on two separate five-point Likert scales ranging from "very good" (5) to "very bad" (1). These two items are included in the Quality from the Patient Perspective questionnaire as two separate questions.
Level of general self-efficacy assessed with the General Self-Efficacy scale | at the date of discharge, an average of 5 days after inclusion
  General self-efficacy measures confidence in one's ability to handle difficult challenges in life. It includes 10 items, which are rated on a four- point Likert scale giving a summary score of 40 for the total scale (10-40).
Quality of care measured with ratings of Medical-technical competence and physical conditions at the ward assessed with the questionnaire Quality from the Patient Perspective. | From date of admission until the date of discharge, up to 60 days of hospitalization.
  The questionnaire comprises four dimension of with the two rational dimensions was used for this specific aim: medical- technical competence (4 items) and physical-technical condition (3 items). Two kinds of assessments are being made at each item: whether things were being done (perceived reality) and whether the right things were being done (subjective significance). For this secondary outcome the assessments of perceived reality is being used. A four-point response scale ranging from 1 (do not agree at all) to 4 (completely agree) forms the basis of ratings, each item also had a response option of "not applicable". Subscales can be reported item by item or combined in a subscale score (average of all responses within the subscale).
Clinical observations of pulse rate | From date of admission until the date of discharge, up to 60 days of hospitalization.
  Frequency of documented pulse rate during hospitalization. The medical records are reviewed retrospectively.
Quality of care assessed as documented information in medical records on current medication at a daily basis and at discharge | From date of admission until the date of the discharge, up to 60 days of hospitalization.
  All information in the medical records during hospitalization are reviewed retrospectively. Rating is made regarding the presence (yes or no) of information on current medication at a daily basis and at discharge.
Quality of care assessed as documented information in medical records on planned medical care at discharge. | From date of admission until the date of discharge, up to 60 days of hospitalization.
  All information in the medical records during hospitalization are reviewed retrospectively. Rating is made regarding the presence (yes or no) of information on planned medical care at discharge.
Clinical observations of weight | From date of admission until date of discharge, up to 60 days of hospitalization.
  Frequency of documented clinical observations of weight (kg) during hospitalization. The medical records are reviewed retrospectively.
Clinical observations of blood pressure | From date of admission until the date of discharge, up to 60 days of hospitalization.
  Frequency of documented clinical observations of systolic and diastolic blood pressure during hospitalization. The medical records are reviewed retrospectively.
Clinical observations of respiratory rate | From date of admission until the date of discharge, up to 60 days of hospitalization.
  Frequency of documented clinical observations of respiratory rate during hospitalization. The medical records are reviewed retrospectively.
Body temperature | From date of admission until the date of discharge, up to 60 days of hospitalization.
  Frequency of documented clinical observations of body temperature (degrees celsius) during hospitalization. The medical records are reviewed retrospectively.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Jakobsson Ung, Associate professor, Principal Investigator — Department of Medicine, Sahlgrenska University Hospital, Gothenburg, Sweden and Institute of Health and Care Sciences, Sahlgrenska Academy at the University of Gothenburg
Locations (1):
- Department of Medicine, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No